CLINICAL TRIAL: NCT03493243
Title: AVAL Cohort Study First Step, Observational Study, After One Year
Brief Title: Teenagers After London Terrorist Attack
Acronym: AVAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Principal Investigator, COULON Nathalie, medical doctor (psychiatrist for children and teenagers), principal Investigator, University Hospital, Brest
Other Study IDs: AVAL (29BRC17.0248)
Record Dates: First submitted 2018-03-20; First posted 2018-04-10 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Adolescent Development; Post Traumatic Stress Disorder; Terrorism
Keywords: Adolescent; Post Traumatic Stress Disorder; Terrorist Attack
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents exposed: Only clinical questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — 2-hour clinical observation

SUMMARY:
* Context: Since March 2012, several terrorist attacks have been perpetrated in France (Toulouse, Montauban, Paris, Nice ...). In March 2017, 53 french teenagers were victims in a terrorist attack in London (Westminster Bridge).
* Main goal = to estimate the psycho-traumatic impact and to describe cares and management of high school students, victims of the terrorist attack in London on 2017, March the 22nd.
* 3 secondary objectives: 1) Clinical (occurrence of Post Traumatic Stress Disorders or other disorders); 2) Epidemiological (risk factors for developing disorders, avoiding care); 3) Preventive and therapeutic.

DETAILED DESCRIPTION:
Inclusion criterion: 53 teenagers of Saint-Joseph high school (Concarneau, France) directly exposed to the terrorist attack.

Methodology: self questionnaires and heterogenous questionnaires; descriptive statistics (means +/- standard deviations; search for a significant difference according to traumatic symptomatology)

ELIGIBILITY:
Inclusion Criteria:

* 53 teenagers, from Concarneau (France) high school, directly exposed from London terrorist attack (22.03.2017).

Exclusion Criteria:

* All persons not directly exposed;
* Relatives of teenagers;
* 3 physically injured teenagers.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * 53 Teenagers;
  * Saint-Joseph high school (29)
  * Directly exposed.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
PTSD | One year after the terrorist attack (Day 1)
  Post Traumatic Stress Disorder (Self-Questionnaire :Posttraumatic stress disorder checklist 5 )

SECONDARY OUTCOMES:
Clinical (occurence of Post Traumatic Stress Disorders or other disorders) | One year after the terrorist attack (Day 1)
  Mini International Neuro-psychiatric Interview for children and adolescent
Epidemiological (risk factors for developing disorders, avoiding care); | One year after the terrorist attack (Day 1)
  LEC = Life Event checklist
Preventive and therapeutic | One year after the terrorist attack (Day 1)
  MINI = Mini International Neuropsychiatric Interview
Epidemiological (risk factors for developing disorders, avoiding care); | One year after the terrorist attack (Day 1)
  ALCES = Adolescent Life Change Event Scale
Epidemiological (risk factors for developing disorders, avoiding care); | One year after the terrorist attack (Day 1)
  EPS 10 = "Echelle de Provisions Sociales Abrégées";
Epidemiological (risk factors for developing disorders, avoiding care); | One year after the terrorist attack (Day 1)
  Whodas 2.0 = World Health Organization Disability Assessment Schedule
Preventive and therapeutic | One year after the terrorist attack (Day 1)
  Questionnaire about use of psychoactive substances

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie V COULON, MD PhD, Study Director — CHU Brest
Locations (2):
- France (2):
  - CHU, Brest
  - HIA Hôpital d'Instruction des Armées Clermont Tonnerre, Brest

IPD SHARING:
Plan to Share IPD: Yes
Secured email aval.france@chu-brest.fr
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: aval.france@chu-brest.fr/

REFERENCES:
- [Derived] Grenon M, Consigny M, Lemey C, Simson JP, Coulon N. Impact of a Terrorist Attack on the Mental Health of Directly Exposed French Adolescents: Study Protocol for the First Step of the AVAL Cohort Study. Front Psychiatry. 2019 Oct 25;10:744. doi: 10.3389/fpsyt.2019.00744. eCollection 2019. PMID 31708812